CLINICAL TRIAL: NCT01604434
Title: Randomized Evaluation of the Use of Plastic Bags to Prevent Neonatal Hypothermia in Developing Countries-Part III
Brief Title: Evaluation of Use of Plastic Bags to Prevent Neonatal Hypothermia-Part III
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no personnel available to enroll in study- decision made to not complete
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Health System, Alabama (Other)
Responsible Party: Principal Investigator, Wally Carlo, Edwin M. Dixon Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 008
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hypothermia
Keywords: Hypothermia; Low birth Weight; Newborn; Incubator; Plastic bag
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incubator-no plastic bag (Sham Comparator): Placement into an incubator without a plastic bag
  Interventions: Procedure: Incubator-no plastic bag
- Incubator-torso bag (Active Comparator): Placement into a plastic bag inside incubator
  Interventions: Procedure: Incubator-torso bag

INTERVENTIONS:
Procedure: Incubator-torso bag — While being placed into an incubator, infant will be placed into a plastic bag to his/her axillae and the bag will be folded and taped to itself to prevent it from covering the infant's nose or mouth. The infant will be wrapped in a blanket over the plastic bag and will receive a cloth hat. He/she will remain in the bag for one hour.
  Arms: Incubator-torso bag
Procedure: Incubator-no plastic bag — Infant will be placed in the incubator, wrapped in a blanket, with a cloth hat, according to standard protocol.
  Arms: Incubator-no plastic bag

SUMMARY:
The overall hypothesis is that plastic bags used in combination with WHO thermoregulation care will reduce the incidence of hypothermia in preterm/low birth weight and full term infants when compared to routine WHO thermoregulation care alone. Part III is for preterm/low birth weight infants with or without a plastic torso wrap during the first hour after birth to assist with temperature regulation during placement in an incubator.

DETAILED DESCRIPTION:
Incubators in the developing world often lack humidifiers. The resting dry heat increases evaporative heat loss, the most prominent form of heat loss in premature infants due to their increased body surface area and immature stratum corneum. By potentially increasing humidity around the infants and decreasing evaporative heat losses, plastic bags may improve incubator warming. This study will compare the incidence of hypothermia in infants placed in an incubator for at least one hour randomized to receive standard incubator protocol (control group) or standard incubator protocol plus a plastic bag covering their torsos and lower extremities (intervention group). The axillary temperature of each infant will be taken before placement into the incubator and one hour later when the bag will be removed. Blood pressure, blood sugar, seizures, weight gain, hyperthermia, death, observation for respiratory distress syndrome, bronchopulmonary dysplasia, pneumothorax, sepsis, intraventricular hemorrhage, periventricular leukomalacia, necrotizing enterocolitis, intestinal perforation, pulmonary hemorrhage, incubator temperature, and humidity, and length of time in an incubator will be recorded throughout the hospitalization for all infants. With an estimated baseline hypothermia rate of 90% and a hypothesized 20% absolute risk reduction (22% relative risk reduction), a sample size of 118 will be used to have a power of 80% and a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Infant admitted to the NICU
* Current weight between 1,000 and 2,500g
* Being placed in an incubator

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Axillary temperature 36.5-37.5 degrees Celsius | 1-72 hours
  Temperature taken per axilla for 1 minute

SECONDARY OUTCOMES:
Blood Pressure | Up to 4 weeks
  Measure of extremity blood pressure per cuff taken during nursery stay
Blood glucose | Up to 4 weeks
  Measure of blood glucose per laboratory value taken per heel stick
Seizure | Up to 4 weeks
  Seizure activity diagnosed by medical doctor or nurse. No electroencephalogram will be done.
Weight gain | Up to 4 weeks
  Infant will be weighed daily and rates of weight gain will be calculated
Respiratory Distress Syndrome (RDS) Respiratory Distress Syndrome (RDS) | Up to 4 weeks
  Documentation of increased work of breathing, retractions, and a need for oxygen, intubation, or surfactant
Bronchopulmonary dysplasia (BPD) | 28 days after birth
  Oxygen requirement at 28 days after birth
Pneumothorax | Up to 4 weeks
  Either chest radiograph documentation or clinical deterioration consistent with air leak
Sepsis | Up to 4 weeks
  Culture proven or culture negative clinically treated course consistent with sepsis
Major brain injury | Up to 4 weeks
  Intracranial hemorrhage grade 3-4 or periventricular leukomalacia documented on cranial ultrasound
Necrotizing enterocolitis or intestinal perforation | Up to 4 weeks
  Documentation of pneumatosis or intestinal perforation on x-ray or treatment course for clinical necrotizing enterocoliities per Bell's Classification stage greater than 1.
Pulmonary hemorrhage | Up to 4 weeks
  Blood seen in the endotracheal tube and treated by physician
Death | Up to 4 weeks
  Cardiorespiratory failure
Hyperthermia | Up to 4 weeks
  Axillary temperature > 38 degrees Celsius per temperature taken per axilla for one minute
Length of time in Incubator | Up to 4 weeks
  Documentation of length of time spent in incubator and number of times placed in incubator
Temperature and humidity | 1 hour
  A recording of the air temperature and humidity within the incubator will be obtained with each axillary temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia